CLINICAL TRIAL: NCT04038632
Title: Impact of an Innovative Childhood TB Diagnostic Approach Decentralized to District Hospital and Primary Health Care Levels on Childhood Tuberculosis Case Detection and Management in High Tuberculosis Incidence Countries
Brief Title: Impact of an Innovative Childhood TB Diagnostic Approach Decentralized to District Hospital and Primary Health Care Levels on Childhood Tuberculosis Case Detection and Management in High Tuberculosis Incidence Countries (TB-Speed Decentralisation)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C18-25
Record Dates: First submitted 2019-06-06; First posted 2019-07-31 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Tuberculosis in Children
Keywords: Decentralized Diagnosis approaches; Childhood TB; Case detection

STUDY DESIGN:
Intervention Model Description: The study will comprise an observation phase, during which there will be no interference with the routine TB childhood diagnosis processes, followed by an intervention phase in participating districts. During the last month of the observation phase, each district will be randomly assigned to implement either DH or PHC focused decentralisation. There will be no individual patient level randomisation.
  The study will also include a nested cohort at both the DH and PHC during the intervention phase for a selected sub-set of children with presumptive TB and all children with a diagnosis of TB who consent to participate. This prospective cohort will enable to further document study endpoints related to follow up (TB treatment outcome) and to document TB diagnosis by assessing spontaneous resolution or resolution under TB treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- District Hospital focused decentralization strategy (Experimental): In this strategy, the patient care level innovative childhood TB diagnostic approach will be implemented at the DH level. PHCs in this district, will only conduct systematic TB screening.
  Interventions: Other: Decentralization of Childhood TB Diagnosis
- Primary Health Center focused decentralization strategy (Experimental): In this strategy, the patient care level innovative childhood TB diagnostic approach will be done at the PHC.
  Interventions: Other: Decentralization of Childhood TB Diagnosis

INTERVENTIONS:
Other: Decentralization of Childhood TB Diagnosis — The patient care level TB diagnostic approach consists of systematic TB screening, clinical evaluation, NPA and stool or sputum testing using Xpert Ultra, and optimised CXR reading will be implemented at DH and PHC levels

SUMMARY:
The TB-Speed Decentralisation study aims to increase childhood Tuberculosis (TB) case detection at district hospital (DH) and Primary health Care (PHC) levels using adapted and child-friendly specimen collection methods, i.e. Nasopharyngeal Aspirate (NPA) and stool samples, sensitive microbiological detection tests (Ultra) close to the point-of-care (Omni/G1(Edge)), reinforced training on clinical diagnosis, and standardized CXR quality and interpretation using digital radiography.

The TB-Speed Decentralisation study will evaluate the impact of an innovative patient care level diagnostic approach deployed at DH and PHC levels, namely the DH focused and the PHC focused decentralization strategies. This is aimed at, improving case detection in 6 high TB incidence in low/moderate resource countries: Cambodia, Cameroon, Côte d'Ivoire, Mozambique, Sierra Leone, and Uganda, and compare effectiveness and cost-effectiveness of the two different decentralization approaches.

The hypothesis is that, in countries with high and very high TB incidence (100-299 and ≥300 cases/100,000 population/year, respectively), a systematic approach to the screening for and diagnosis of TB in sick children presenting to the health system will increase childhood TB case detection, especially PTB, which represents the majority of the disease burden (>75% of case). The study also hypothesizes that sputum collection using battery-operated suction machines and microbiological TB diagnosis using Omni/G1 (Edge) can be decentralized to PHC level, thus enabling TB diagnosis and treatment in children at PHC level.

DETAILED DESCRIPTION:
This will be an operational research study using:

* a before and after cross-sectional design to assess the impact of decentralizing an innovative childhood TB diagnostic approach
* a cross-sectional and nested cohort design to compare two different decentralization strategies at DH and PHC levels.
* quantitative and qualitative methods The intervention will be at two levels: at patient care level where an innovative childhood TB diagnostic approach will be implemented, and at health systems level where two distinct decentralization strategies will be implemented. The patient care level TB diagnostic approach consists of systematic TB screening, clinical evaluation, NPA and stool or sputum testing using Xpert Ultra, and optimised CXR reading. The two decentralization strategies are the DH-focused and the PHC-focused implementation of the innovative childhood TB diagnostic approach. Two districts per participating countries will be randomly assigned to implement the DH or PHC-focused strategies.

The study will also include a nested cohort at both the DH and PHC during the intervention phase for a selected sub-set of children with presumptive TB and all children with a diagnosis of TB that consent to participate. This prospective cohort will enable to further document study endpoints related to follow up (TB treatment outcome) and to document TB diagnosis by assessing spontaneous resolution or resolution under TB treatment.

The study will comprise an observation phase followed by an intervention phase in participating districts. During the last month of the observation phase, each district will be randomly assigned to implement either DH or PHC-focused decentralisation. There will be no patient level randomisation.

During this 3-month observation phase, the study will 1) describe the childhood TB diagnosis data and practices; 2) describe the referral processes and outcomes of referrals for TB diagnosis and treatment where feasible and 3) assess existing challenges in childhood TB diagnosis and treatment, as well as readiness (including potential challenges) for the study intervention implementation. There will be no interference with the routine TB childhood diagnosis processes.

Mixed-methods (quantitative and qualitative) will be used including the collection of retrospective and prospective aggregated data by study nurses from facility registers, the implementation of a self-administered questionnaire among all healthcare workers (HCWs), the observation of consultations and care provided, and the conduct of individual interviews with HCWs and key informants.

At the beginning of the intervention phase, a 3-months preparation period will set up the health facilities for decentralization by providing equipment, materials, and reagents, training health workers in childhood TB care, in NPA and stool collection and testing on Ultra, setting up G1 (Edge) at PHC or G4 at DH if not already available and digital CXR and CXR quality control. Existing health care workers will be trained in childhood TB care according to the National Tuberculosis Program (NTP) guidelines, and also in NPA and stool collection and testing on Ultra for study purposes.

Implementation of the innovative childhood TB diagnostic approach at the selected DH and PHC will start as soon as sites are equipped and HCWs trained in childhood TB care and NPA and stool collection, and will implement continued capacity building at sites, regular clinical mentoring visits with NTP or their representative, and continued CXR quality control.

The 6-month prospective cohort follow-up study will be initiated immediately and will consecutively include every tenth child with presumptive TB and all children diagnosed with TB.

Individual data collection will be initiated as soon as the innovative childhood TB diagnostic approach including NPA and stool sample collection and Ultra testing is implemented in the site and will be conducted throughout the intervention phase to document secondary endpoints. Aggregated data for TB screening will be collected throughout the study.

Feasibility, acceptability, and compliance to the intervention protocol will be assessed by mixed methods including a repeat self-administered questionnaire among all HCWs, observations of consultations and care provided, and individual interviews with HCWs, National TB program & local health authorities representatives, and beneficiaries. i.e. parents/guardians.

ELIGIBILITY:
Inclusion Criteria:

* Sick children seeking care at Oupatient Department of District Hospital or Primary Health Center
* Age <15 years

Exclusion Criteria:

- None

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3106 (Actual)
Dates: Start 2020-03-07 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Children diagnosed with TB | Day 0
  Proportion of TB cases detected among sick children routinely attending outpatient services before and after the intervention

SECONDARY OUTCOMES:
TB case detection | Month 6
  Proportion of TB cases (confirmed and unconfirmed) detected among children identified as presumptive TB
TB screening in outpatient children - 1 | Day 7
  Proportion of children screened for TB among sick children attending outpatient services
TB screening in outpatient children - 2 | Day 7
  Proportion of children identified with presumptive TB among children screened
Feasibility of implementing the different diagnostic approach components - 1 | Day 7
  Proportion of children with presumptive TB enrolled in the study receiving the different components of the innovative childhood TB diagnostic approach (NPA and stool or sputum sampling attempt and success, sample testing with Ultra and results, clinical evaluation, CXR and interpretation, full diagnostic package)
Feasibility of implementing the different diagnostic approach components - 2 | Day 7
  Time to sample test and results delivery to clinician
Feasibility of implementing the different diagnostic approach components - 3 | Day 7
  Number of visits to the health facility until final diagnosis
TB treatment uptake and time to TB treatment initiation - 1 | Month 6
  Proportion of children initiating TB treatment among those diagnosed as TB
TB treatment uptake and time to TB treatment initiation - 2 | Month 6
  Time from positive TB screening to TB treatment initiation
Cost-effectiveness from the health services perspective | Month 22
  Incremental-Cost Effectiveness Ratio (ICER) of the diagnostic approach
Acceptability by health care providers, NTPs and health authorities, and beneficiaries | Day 0
  Perceptions and experience of the intervention by healthcare workers (HCWs), the NTP and health authorities, and the beneficiaries (parents/guardians)
Fidelity of the implementation of the diagnostic approach as compared to the protocol and study procedures - 1 | Month 6
  Changes in the intervention implementation as compared to 1) study standard implementation procedures and 2) country implementation procedures.
  These changes could be related to NTP guidelines dispositions, adaptation to local context and constraints not initially planned per standard and country implementation procedures
Fidelity of the implementation of the diagnostic approach as compared to the protocol and study procedures - 2 | Month 22
  Proportion of clinical mentoring visits performed per study procedures; proportion of health facilities implementing NPA and stool sample collection and performing sample processing and Ultra testing per study procedures
Performance of the diagnostic approach at patient level | Month 6
  Sensitivity and specificity of the diagnostic approach as compared to the reference diagnosis based on the Case Definitions for Classification of Intrathoracic Tuberculosis in Children for clinical research
TB treatment outcome | Month 6
  TB treatment outcome as defined by WHO
Diagnostic performance of CXR reading by clinicians at DH and PHC levels | Month 6
  Sensitivity and specificity of CXR reading by clinicians at DH and PHC to detect lesions suggestive of TB as compared to the reference reading (independent reading by external radiologist experts)
Added value of CXR in the diagnosis of TB in children as compared to microbiology and clinical evaluation only | Month 6
  Proportion of children diagnosed with TB based on CXR and incremental yield of TB detection with CXR results as compared to microbiological (Ultra on NPA and stool or sputum) and clinical evaluation, respectively
Uptake of the quality control of the CXR reading | Month 6
  Proportion of CXR selected for quality review assessed by the reference reviewer and time to results of the quality control to the clinic

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Marcy, PhD, Principal Investigator — University of Bordeaux; Maryline Bonnet, PhD, Principal Investigator — Institut de Recherche pour le Developpement; Eric Wobudeya, PhD, Principal Investigator — MU-JHU Care Ltd
Locations (59):
- Cambodia (10):
  - Angroka Rh, Angroka
  - Taphem Hc, Angroka
  - Tropang Andert Hc, Angroka
  - Batheay Rh, Batheay
  - Choeung Chnok Hc, Batheay
  - Tumnub Hc, Batheay
  - Nhaeng Nhang Hc, Nhaeng Nhang
  - KUS HC, Phumĭ Kŭs
  - Phaav HC, Ph’av
  - Sambour Hc, Sambour
- Cameroon (10):
  - Csi Messngssang, Bafia
  - HD BAFIA, Bafia
  - Csi Balamba Bafia, Balamba
  - Cma Batchenga, Batchenga
  - Cma Bokito Bafia, Bokito
  - Csi Essong, Essong
  - Cma Kiiki Bafia, Kiiki
  - Cma Fomakap, Obala
  - Csi Ngogo, Obala
  - Obala Hosp, Obala
- Côte d’Ivoire (10):
  - Dr Banteapleu, Banteapleu
  - Csu Dakpadou, Dakpadou
  - Csr Daleu, Daleu
  - H G de Danane, Danané
  - Csu Kouan-Houle, Kouan Houlé
  - Csu Mahapleu, Mahapleu
  - Csr Medon, Médon
  - CMS SAGO, Sago
  - Dr de Sahoua, Sahoua
  - H G Sassandra, Sassandra
- Mozambique (9):
  - Chiaquelane, Chiaquelane
  - Chibonzane, Chibonzane
  - Chidenguele, Chidenguele
  - Chalocuane, Chokwé
  - HOKWE, Chokwé
  - Hosp Rural Chokwe, Chokwé
  - MACUACUA, Macuácua
  - Hospital Rural de Manjacaze, Manjacaze
  - Laranjeira, Manjacaze
- Sierra Leone (10):
  - Babara Chc, Babara
  - Bo Govt Hosp, Bo
  - New Police barracks, Bo
  - Gbinti Chc, Gbinti
  - Gerihun Chc, Gerihun
  - Koribondo Chc, Koribondo
  - Mange Chc, Mange
  - Njala University Chc, Njala
  - Petifu Chc, Petifu
  - Port Loko Govt Hosp, Port Loko
- Uganda (10):
  - Buyamba Hc Iii, Buyamba
  - Kambuga Hospital, Kambuga
  - Kanungu Hciv, Kanungu
  - Kanyantorogo Hciii, Kanyantorogo
  - Lwamaggwa Hc Iii, Lwamaggwa
  - Lwanda Hc Iii, Lwanda
  - St Bernards Manya Hc Iii, Manya
  - Matanda Hciii, Matanda
  - Nyamirama HC III, Nyamirama
  - Rakai Hospital, Rakai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi B, De Lima YV, Massom DM, Kaing S, Banga MF, Kamara ET, Sesay S, Borand L, Taguebue JV, Moh R, Khosa C, Breton G, Mwanga-Amumpaire J, Bonnet M, Wobudeya E, Marcy O, Orne-Gliemann J; TB-Speed Decentralization study group. Acceptability of decentralizing childhood tuberculosis diagnosis in low-income countries with high tuberculosis incidence: Experiences and perceptions from health care workers in Sub-Saharan Africa and South-East Asia. PLOS Glob Public Health. 2023 Oct 11;3(10):e0001525. doi: 10.1371/journal.pgph.0001525. eCollection 2023. PMID 37819919
- [Derived] d'Elbee M, Harker M, Mafirakureva N, Nanfuka M, Huyen Ton Nu Nguyet M, Taguebue JV, Moh R, Khosa C, Mustapha A, Mwanga-Amumpere J, Borand L, Nolna SK, Komena E, Cumbe S, Mugisha J, Natukunda N, Mao TE, Wittwer J, Benard A, Bernard T, Sohn H, Bonnet M, Wobudeya E, Marcy O, Dodd PJ; TB-Speed Health Economics Study Group. Cost-effectiveness and budget impact of decentralising childhood tuberculosis diagnosis in six high tuberculosis incidence countries: a mathematical modelling study. EClinicalMedicine. 2024 Mar 21;70:102528. doi: 10.1016/j.eclinm.2024.102528. eCollection 2024 Apr. PMID 38685930
- [Derived] Wobudeya E, Nanfuka M, Ton Nu Nguyet MH, Taguebue JV, Moh R, Breton G, Khosa C, Borand L, Mwanga-Amumpaire J, Mustapha A, Nolna SK, Komena E, Mugisha JR, Natukunda N, Dim B, de Lauzanne A, Cumbe S, Balestre E, Poublan J, Lounnas M, Ngu E, Joshi B, Norval PY, Terquiem EL, Turyahabwe S, Foray L, Sidibe S, Albert KK, Manhica I, Sekadde M, Detjen A, Verkuijl S, Mao TE, Orne-Gliemann J, Bonnet M, Marcy O; TB-Speed Decentralisation study group. Effect of decentralising childhood tuberculosis diagnosis to primary health centre versus district hospital levels on disease detection in children from six high tuberculosis incidence countries: an operational research, pre-post intervention study. EClinicalMedicine. 2024 Mar 21;70:102527. doi: 10.1016/j.eclinm.2024.102527. eCollection 2024 Apr. PMID 38685921
- See also: TB-Speed project official website — http://www.tb-speed.com